CLINICAL TRIAL: NCT04756271
Title: Safety and Immunogenicity of Oxford AstraZeneca Vaccine in Zagazig University Hospital Health-care Workers
Brief Title: Safety and Immunogenicity of Oxford AstraZeneca Vaccine Against COVID-19 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Noha M Hammad, MD, Principal investigator, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6738-14-2-21
Record Dates: First submitted 2021-02-13; First posted 2021-02-16 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Vaccine Adverse Reaction; Seroconversion
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health-care workers (Experimental): Healthy health-care workers at Zagazig University Hospital who opt by their free well to administer 2 doses of SARS-Cov-2 inactivated vaccine at 0 and 21 days. Blood samples will be withdrawn from them to investigate the immune response to the given vaccine
  Interventions: Biological: SARS-Cov-2 neutralizing antibody titer

INTERVENTIONS:
Biological: SARS-Cov-2 neutralizing antibody titer — Quantitation of SARS-Cov-2 antibody titer at baseline after each dose of the vaccine

SUMMARY:
After SARS-COV-2 inactivated vaccine authorization for use in different countries including Egypt, investigating its immunogenicity, safety, and efficacy in preventing COVID-19 infection is highly needed. In Egypt, immunization of HCWs in isolation hospitals by SARS-COV-2 inactivated vaccine is now a national priority. Moreover, data and reports regarding the application of vaccine are still limited and deficient.

DETAILED DESCRIPTION:
This study will be conducted at Zagazig University hospital. Laboratory work will be implemented at Immunology Research Laboratory at Microbiology and Immunology Department, Faculty of Medicine, Zagazig University. A representative sample will be drawn from healthcare workers (HCWs) at Zagazig University Hospital. Assessment of inclusion and exclusion criteria by history taking. Blood samples will be drawn from HCWs by direct venipuncture before the start of immunization and 14 days after immunization. The incidence of any adverse reactions after each immunization will be recorded. SARS-CoV-2 neutralizing antibodies will be detected by enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

-Healthy healthcare workers

Exclusion Criteria:

* Healthy healthcare workers' refusal.
* Pregnancy and lactation.
* Confirmed acute cases of SARS-CoV-2 Infection
* Having a history of SARS-CoV-2 infection in the past 3 months.
* Fever (body temperature > 37.0 ℃), dry cough, fatigue, nasal obstruction, runny nose, pharyngeal pain, myalgia, diarrhea, shortness of breath and dyspnea occurred within 14 days before vaccination.
* History of allergy to any vaccines
* Previous vaccination within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 7 days after each dose
  Incidence of adverse reactions after each dose of the vaccine
Seroconversion rate of neutralizing antibody | 84 days after each dose
  Neutralizing antibody assay will be performed after each dose of the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Noha M Hammad, MD, Principal Investigator — Faculty of Medicine, Zagazig University , Zagazig, Egypt
Locations (1):
- Zagazig University Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No